CLINICAL TRIAL: NCT02705040
Title: Roles of microRNAs in the Development of Osteoporosis in Men - Preliminary Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TMU-JIRB 201310015
Record Dates: First submitted 2016-01-29; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-01

CONDITIONS: Osteoporosis
Keywords: male osteoporosis; miRNA; biomarker
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal: bone mineral density T>=-1.0
  Interventions: Other: Osteopenia; Other: Osteoporosis
- Osteopenia: bone mineral density -1.0>T>=-2.5
  Interventions: Other: Normal; Other: Osteoporosis
- Osteoporosis: bone mineral density T<-2.5
  Interventions: Other: Normal; Other: Osteopenia

INTERVENTIONS:
Other: Normal — bone mineral density T>=-1.0
  Groups: Osteopenia; Osteoporosis
Other: Osteopenia — bone mineral density -1.0>T>=-2.5
  Groups: Normal; Osteoporosis
Other: Osteoporosis — bone mineral density T<-2.5
  Groups: Normal; Osteopenia

SUMMARY:
This study is aimed to evaluate the roles of specific miRNAs in osteoporosis in men.

DETAILED DESCRIPTION:
In the past, osteoporosis is usually viewed as a woman disease. However, men and women are shown to lose their bone mass at the same rate by more than 65 of age, and osteoporosis in men causes higher mortality in men than those in women. Thus, osteoporosis in men has recently aroused public attention. Androgen deficiency was the main cause leading to osteoporosis. Bone structure is maintained by a dynamic balance of osteoblast-mediated bone formation and osteoclast-mediated bone resorption. Androgens and androgen receptor (AR) play critical roles in regulation of bone formation and resorption. MicroRNAs (miRNAs) are non-coding small RNAs and participate in regulating activities of osteoblasts and osteoclasts by postranslationally targeting certain gene expressions. miR-133 and -135 can target BMP-2, Runx2, and Smad5 and then regulate osteoblast differentiation. Likewise, miR-141 and -200a negatively regulated osteoblast differentiation. Nevertheless, the functional roles of miRNAs in osteoporosis in men are still unknown. In addition, miRNA are stable and can be detected in the blood as novel biomarkers for certain diseases. A recent study analyzed the levels of miRNAs in circulating monocytes of 10 high and 10 low bone mineral density postmenopausal Caucasian women and found miR-133a is a potential biomarker for postmenopausal osteoporosis. In comparison, the roles of blood miRNAs in osteoporosis in men have not been evaluated. Therefore, this study is aimed to evaluate the roles of specific miRNAs in osteoporosis in men.

ELIGIBILITY:
Inclusion Criteria:

1. Twenty oriental men (mean age, 80 years; age range, 70-90 years).
2. Candidates have no clinical evidence or history of focal lesions of the femur; previous hip surgery or irradiation; hip trauma; spinal trauma.
3. Participants who have thoroughly understood and signed the consent form.
4. Ten normal adult male (age range, 20-40 years).

Exclusion Criteria:

1. Participants with secondary causes of osteoporosis, such as thyroid, parathyroid disease, osteogenesis imperfect and osteomalacia.
2. Participants with Paget's disease, serious liver disease, serious renal disease (indicated by a serum creatinine concentration of more than 1.6mg/dL).
3. Participants who currently or have history of using steroids or hormone replacement therapy.
4. Participants who fail to sign to the consent form.

Ages: 70 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The oriental men
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 30 minutes
  T scale

CONTACTS AND LOCATIONS:
Overall Officials: Ruei-Ming Chen, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University Wanfang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No